CLINICAL TRIAL: NCT06560203
Title: Safety and Efficacy of Endovascular Treatment for Acute Basilar Artery Occlusion in the Extended Time Window -a Prospective, Multicenter, Randomized Controlled, Open-label Clinical Trial
Brief Title: Basilar Artery Occlusion Chinese Endovascular Trial in the Extended Time Window
Acronym: BAOCHE2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAOCHE-2
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Ischemic Stroke; Basilar Artery Occlusion
Keywords: Mechanical thrombectomy; Extended time window
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mechanical thrombectomy group (Experimental): Researchers can choose to deal with the stenosis or occlusion of blood vessels according to their own judgment, including stent thrombectomy, thrombus aspiration, balloon angioplasty, stent replacement, intra-arterial thrombolysis or various combinations of these methods.
  Interventions: Procedure: Mechanical thrombectomy
- best medical management agroup (No Intervention): Best Medical Treatment and maximum supportive care according to local guidelines, not including mechanical thrombectomy, no intra-arterial treatment.

INTERVENTIONS:
Procedure: Mechanical thrombectomy — Neurointerventionist determine whether to proceed with interventional therapy after assessing the location and degree of occlusion, the tortuosity of the access vessel, and the presence of stenosis or occlusion in the proximal artery. In cases where there is no proximal stenosis or occlusion, mechanical thrombectomy is performed, and the specific thrombectomy strategy is tailored by the researcher based on the patient's condition. For lesions associated with proximal vascular stenosis or occlusion, it is necessary to navigate the catheter through the proximal stenosis or occlusion to access the intracranial occlusion. Researchers have the discretion to treat the stenotic or occluded vessels, which may include options such as no treatment, stent thrombectomy, thrombus aspiration, balloon angioplasty, stent replacement, intra-arterial thrombolysis or various combinations of these methods.
  Arms: mechanical thrombectomy group

SUMMARY:
A prospective, multi-center, randomized, controlled, open-label, blinded-endpoint trial to evaluate the safety and efficacy of endovascular mechanical thrombectomy for acute basilar artery occlusion in the extended time window

DETAILED DESCRIPTION:
This trial aims to evaluate the hypothesis that mechanical thrombectomy is superior to medical management alone in achieving favorable outcomes in subjects presenting with stroke due to basilar artery occlusion in the extended time window of 24-72 hours from symptom onset or time last seen well. In this trial, the randomization will employ a 2:1 ratio of mechanical thrombectomy versus best medical management alone. Randomization will be stratified according to age (18-70 or >70), baseline NIHSS (6-20 or >20) and therapeutic window (24-48 hours or >48 hours). For the primary endpoint, subjects will be followed for 90 days post-randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Posterior circulation acute ischemic stroke within 24-72 hours from symptom onset/last seen well (except for isolated vertigo), where patient is ineligible for IV thrombolytic treatment or the treatment is contraindicated (e.g., patient presents beyond recommended time from symptom onset), or where patient has received IV thrombolytic therapy without recanalization.
2. Occlusion (TIMI 0-1) of the basilar artery or intracranial segments of both vertebral arteries (V4) as evidenced by CTA/MRA/DSA.
3. Age ≥18 and ≤ 80.
4. Baseline NIHSS score obtained prior to randomization must be equal or higher than 6 points.
5. No significant pre-stroke functional disability (mRS ≤ 1).
6. Patient treatable within 72 hours of symptom onset. Symptom onset is defined as the point in time the patient was last seen well (at baseline) if patients are unable to provide a reliable history or the point in time when symptoms have started if patients can provide a reliable history.
7. Informed consent obtained from patient or authorized patient surrogate

Exclusion Criteria:

Clinical criteria

1. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 3.0.
2. Baseline platelet count < 50000/µL.
3. Baseline blood glucose of < 50mg/dL or >400mg/dl.
4. Severe, sustained hypertension (SBP > 220 mm Hg or DBP > 110 mm Hg) NOTE: If the blood pressure can be successfully reduced and maintained below these levels using commonly used medications in China for these purposes (including iv antihypertensive drips), the patient can be enrolled.
5. Patients in whom baseline NIHSS can not be obtained by a neurologist or emergency physician prior to sedation or intubation.
6. Seizures at stroke onset which would preclude obtaining a baseline NIHSS.
7. Serious, advanced, or terminal illness with anticipated life expectancy of less than one year.
8. History of life threatening allergy (more than rash) to contrast medium.
9. Patients with acute stroke within the first 48 hours after percutaneous cardiac, cerebrovascular interventions and major surgery .
10. Renal insufficiency with creatinine ≥ 3 mg/dl.
11. Woman of childbearing potential who is known to be pregnant or lactating or who has a positive pregnancy test on admission.
12. Subject participating in a study involving an investigational drug or device that would impact this study.
13. Known diagnosis or clinical suspicion of cerebral vasculitis.
14. Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations. This excludes patients who are severely demented, require constant assistance in a nursing home type setting or who live at home but are not fully independent in activities of daily living (toileting, dressing, eating, cooking and preparing meals, etc.).
15. Unlikely to be available for 90 days follow-up (e.g. no fixed home address, visitor from overseas).
16. Any other condition that, in the opinion of the investigator will pose a significant hazard to the subject if participating in the trial.

    Neuroimaging criteria
17. Hypodensity with a posterior circulation Acute Stroke Prognosis Early CT score (pc-ASPECTS) < 6 and Pons-midbrain-index of ≥ 3 on CT angiography source images or MR with diffusion-weighted imaging or non-contrast CT.
18. CT or MR evidence of hemorrhage (the presence of microbleeds on MRI is allowed).
19. Complete cerebellar infarct on CT or MRI with significant mass effect and compression of the fourth ventricle.
20. Complete bilateral thalamic infarction on CT or MRI.
21. Evidence of vertebral occlusion, high grade stenosis or arterial dissection in the extracranial or intracranial segment that cannot be treated or will prevent access to the intracranial clot or excessive tortuosity of cervical vessels precluding device delivery/deployment.
22. Subjects with occlusions in both anterior and posterior circulation.
23. Evidence of intracranial tumor (except small meningioma).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in proportion of patients achieving favorable outcomes (defined as mRS 0-3) at 90 days | 90 days
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])

SECONDARY OUTCOMES:
Dramatic early favorable response | 24 (-2/+12) hours
  Dramatic early favorable response as determined by an National Institute of Health stroke scale (NIHSS) of 0-2 or NIHSS improvement ≥ 8 points at 24 (-2/+12) hours.
Dichotomized mRS score (0-2 versus 3-6 ) | 90 days
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])
Ordinal Shift analysis of mRS at 90 days | 90 days
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])
Barthel Index at 90 days | 90 days
  An ordinal scale which measures a person's ability to complete activities of daily living (ADL).
Quality of life analysis as measured by EuroQol Five Dimensions (EuroQol/EQ-5D) | 90 days
  EuroQol Five Dimensions (EuroQol/EQ-5D) is a well-known and widely used health status instrument, and could be used to measure, compare and value health status across disease areas.
Difference in proportion of patients with mRS 0-2 scores between the two groups at 12 months. | 12 months
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])
Difference in proportion of patients with mRS 0-3 scores between the two groups at 12 months. | 12 months
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])
Proportion of basilar artery recanalization | 24-72 hours (both treatment groups); post procedure immediately (thrombectomy arm)
  Vessel recanalization evaluated by CT angiography (CTA), MR Angiography (MRA) or conventional angiography at 24-72 hours in both treatment groups assessed by Arterial Occlusive Lesion（AOL) grades and adjudicated by a central core-lab.
  Vessel recanalization post procedure in the thrombectomy arm assessed by mTICI grades. Successful recanalization is defined as mTICI (Modified Thrombolysis in Cerebral Infarction) 2b or 3 on the post-procedure angiogram.

OTHER OUTCOMES:
Mortality | 90 days
  Death
Symptomatic intracranial hemorrhage | 24-72 hours
  Clinically significant ICH rates at 24-72 hours. All intracerebral hemorrhages will be classified by a central core-lab using the Heidelberg criteria. Symptomatic intracranial hemorrhage will be defined as per the following definition: deterioration in NIHSS score of ≥ 4 points and evidence of intraparenchymal hemorrhage type 2 in the 24 to 72 hours follow-up imaging scans.
Serious adverse events (SAE) | 90 days, 12 months, during follow-up
  All SAE during follow-up in all randomized patients.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The study is proceeding.

REFERENCES:
- [Result] Jovin TG, Li C, Wu L, Wu C, Chen J, Jiang C, Shi Z, Gao Z, Song C, Chen W, Peng Y, Yao C, Wei M, Li T, Wei L, Xiao G, Yang H, Ren M, Duan J, Liu X, Yang Q, Liu Y, Zhu Q, Shi W, Zhu Q, Li X, Guo Z, Yang Q, Hou C, Zhao W, Ma Q, Zhang Y, Jiao L, Zhang H, Liebeskind DS, Liang H, Jadhav AP, Wen C, Brown S, Zhu L, Ye H, Ribo M, Chang M, Song H, Chen J, Ji X; BAOCHE Investigators. Trial of Thrombectomy 6 to 24 Hours after Stroke Due to Basilar-Artery Occlusion. N Engl J Med. 2022 Oct 13;387(15):1373-1384. doi: 10.1056/NEJMoa2207576. PMID 36239645
- [Result] Tao C, Nogueira RG, Zhu Y, Sun J, Han H, Yuan G, Wen C, Zhou P, Chen W, Zeng G, Li Y, Ma Z, Yu C, Su J, Zhou Z, Chen Z, Liao G, Sun Y, Ren Y, Zhang H, Chen J, Yue X, Xiao G, Wang L, Liu R, Liu W, Liu Y, Wang L, Zhang C, Liu T, Song J, Li R, Xu P, Yin Y, Wang G, Baxter B, Qureshi AI, Liu X, Hu W; ATTENTION Investigators. Trial of Endovascular Treatment of Acute Basilar-Artery Occlusion. N Engl J Med. 2022 Oct 13;387(15):1361-1372. doi: 10.1056/NEJMoa2206317. PMID 36239644
- [Result] Kobeissi H, Ghozy S, Adusumilli G, Kadirvel R, Brinjikji W, Rabinstein AA, Kallmes DF. Endovascular Therapy for Stroke Presenting Beyond 24 Hours: A Systematic Review and Meta-analysis. JAMA Netw Open. 2023 May 1;6(5):e2311768. doi: 10.1001/jamanetworkopen.2023.11768. PMID 37140919
- [Result] Purrucker JC, Ringleb PA, Seker F, Potreck A, Nagel S, Schonenberger S, Berberich A, Neuberger U, Mohlenbruch M, Weyland C. Leaving the day behind: endovascular therapy beyond 24 h in acute stroke of the anterior and posterior circulation. Ther Adv Neurol Disord. 2022 May 25;15:17562864221101083. doi: 10.1177/17562864221101083. eCollection 2022. PMID 35646160
- [Result] Pandhi A, Chandra R, Abdulrazzak MA, Alrohimi A, Mahapatra A, Bain M, Moore N, Hussain MS, Bullen J, Toth G. Mechanical thrombectomy for acute large vessel occlusion stroke beyond 24 h. J Neurol Sci. 2023 Apr 15;447:120594. doi: 10.1016/j.jns.2023.120594. Epub 2023 Mar 2. PMID 36893513
- [Result] Markus HS. Reperfusion therapy for stroke: From improving global access, to thrombectomy beyond 24 hours. Int J Stroke. 2024 Mar;19(3):248-250. doi: 10.1177/17474930241232131. No abstract available. PMID 38420839
- [Result] Dhillon PS, Butt W, Podlasek A, Barrett E, McConachie N, Lenthall R, Nair S, Malik L, James MA, Dineen RA, England TJ. Endovascular thrombectomy beyond 24 hours from ischemic stroke onset: a propensity score matched cohort study. J Neurointerv Surg. 2023 Mar;15(3):233-237. doi: 10.1136/neurintsurg-2021-018591. Epub 2022 Feb 15. PMID 35169031
- [Result] Rodriguez-Calienes A, Galecio-Castillo M, Vivanco-Suarez J, Mohamed GA, Toth G, Sarraj A, Pujara D, Chowdhury AA, Farooqui M, Ghannam M, Samaniego EA, Jovin TG, Ortega-Gutierrez S. Endovascular thrombectomy beyond 24 hours from last known well: a systematic review with meta-analysis. J Neurointerv Surg. 2024 Jun 17;16(7):670-676. doi: 10.1136/jnis-2023-020443. PMID 37355251
- [Result] Shaban A, Al Kasab S, Chalhoub RM, Bass E, Maier I, Psychogios MN, Alawieh A, Wolfe SQ, Arthur AS, Dumont TM, Kan P, Kim JT, De Leacy R, Osbun JW, Rai AT, Jabbour P, Park MS, Crosa RJ, Mascitelli JR, Levitt MR, Polifka AJ, Casagrande W, Yoshimura S, Matouk C, Williamson R, Gory B, Mokin M, Fragata I, Romano DG, Chowdhry SA, Moss M, Behme D, Limaye K, Spiotta AM, Samaniego EA. Mechanical thrombectomy for large vessel occlusion strokes beyond 24 hours. J Neurointerv Surg. 2023 Dec 21;15(e3):e331-e336. doi: 10.1136/jnis-2022-019372. PMID 36593118
- [Result] Liu S, Cao W, Wu L, Wen A, Zhou Y, Xiang Z, Rao W, Yao D. Endovascular treatment over 24 hours after ischemic stroke onset: a single-center retrospective study. Neuroradiology. 2023 Apr;65(4):793-804. doi: 10.1007/s00234-022-03105-6. Epub 2022 Dec 23. PMID 36550266
- [Result] Mohamed GA, Nogueira RG, Essibayi MA, Aboul-Nour H, Mohammaden M, Haussen DC, Ruiz AM, Gross BA, Kuybu O, Salem MM, Burkhardt JK, Jankowitz B, Siegler JE, Patel P, Hester T, Ortega-Gutierrez S, Farooqui M, Galecio-Castillo M, Nguyen TN, Abdalkader M, Klein P, Charles JH, Saini V, Yavagal DR, Jumah A, Alaraj A, Peng S, Hafeez M, Tanweer O, Kan P, Scaggiante J, Matsoukas S, Fifi JT, Mayer SA, Chebl AB. Tissue Clock Beyond Time Clock: Endovascular Thrombectomy for Patients With Large Vessel Occlusion Stroke Beyond 24 Hours. J Stroke. 2023 May;25(2):282-290. doi: 10.5853/jos.2023.00017. Epub 2023 May 30. PMID 37282375
- [Result] Sarraj A, Mlynash M, Heit J, Pujara D, Lansberg M, Marks M, Albers GW. Clinical Outcomes and Identification of Patients With Persistent Penumbral Profiles Beyond 24 Hours From Last Known Well: Analysis From DEFUSE 3. Stroke. 2021 Mar;52(3):838-849. doi: 10.1161/STROKEAHA.120.031147. Epub 2021 Feb 10. PMID 33563012
- [Result] Christensen S, Mlynash M, Kemp S, Yennu A, Heit JJ, Marks MP, Lansberg MG, Albers GW. Persistent Target Mismatch Profile >24 Hours After Stroke Onset in DEFUSE 3. Stroke. 2019 Mar;50(3):754-757. doi: 10.1161/STROKEAHA.118.023392. PMID 30735466